CLINICAL TRIAL: NCT05471778
Title: The Effect of Postoperative Music and Comedy Movie Application on Surgical Pain and Kinesiophobia After Total Knee Artroplasty
Brief Title: Effects of Music and Comedy Application on Pain and Kinesyophobia in Patients With TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malatya Turgut Ozal University (Other)
Responsible Party: Principal Investigator, Gurkan KAPIKIRAN, Assistant Professor, Malatya Turgut Ozal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021-178
Record Dates: First submitted 2022-07-19; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Arthroplasty Complications; Kinesiophobia
Keywords: Music; Comedy movie; Kinesiophobia; Pain; Total knee arthroplasty
MeSH Terms: conditions — Kinesiophobia; Pain

STUDY DESIGN:
Intervention Model Description: This study was conducted as a randomized controlled trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- comedy movie group (Experimental): Sociodemographic information form, kinesiophobia scale and numerical pain scale were administered to the patients in the comedy group on the first evening after surgery. 25-minute comedy film was watched. Afterwards, the kinesiophobia scale and the numerical pain scale were applied again.
  Interventions: Behavioral: Watching comedy movie
- Music group (Experimental): Sociodemographic information form, kinesiophobia scale and numerical pain scale were administered to the patients in the music group on the first evening after surgery. 25 minutes of music (nature sound) was played. Afterwards, the kinesiophobia scale and the numerical pain scale were applied again.
  Interventions: Behavioral: listening to music
- Control group (No Intervention): In the follow-up of the patient, no application was made other than clinical protocols. Sociodemographic information form, kinesiophobia scale and numerical pain scale were administered to the patients in the control group on the first evening after surgery. No intervention was made. Afterwards, the kinesiophobia scale and the numerical pain scale were applied again.

INTERVENTIONS:
Behavioral: Watching comedy movie — A 25-minute comedy film created by the researchers was watched.
  Arms: comedy movie group
Behavioral: listening to music — 25 minutes of music created by the researchers was played.
  Arms: Music group

SUMMARY:
Total knee arthroplasty (TKA) is a surgical procedure used to restore painless joint function and increase patients' activities of daily living in patients with progressive knee osteoarthrosis. Kinesiophobia can be seen in patients suffering from pain. It is stated that the incidence of kinesiophobia in TKA patients is 24.4%. Based on this information, this study was planned.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a surgical procedure used to restore painless joint function and increase patients' activities of daily living in patients with progressive knee osteoarthrosis. Kinesiophobia can be seen in patients suffering from pain. It is stated that the incidence of kinesiophobia in TKA patients is 24.4%. Pain etc. While conditions can be relieved by pharmacological treatment methods, non-pharmacological treatments can be effective in relieving patients' pain. With the relief of pain, it will be possible to eliminate the kinesiophobia experienced by the patients. It is known that humor, which is among the non-pharmacological treatment methods, increases the pain resistance of the patients, reduces the stress hormone, and strengthens the immune system. It is reported in the literature that listening to music, another non-pharmacological treatment, is also effective in relieving pain after TKA. For this reason, the study was planned to determine the effect of postoperative music and comedy films on kinesiophobia and pain in patients undergoing TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who agreed to participate in the study,
* Patients undergoing TKA
* Patients without a disabling psychiatric disorder

Exclusion Criteria:

* Patients under the age of 18 who do not agree to participate in the study.
* Those who have a psychiatric diagnosis that prevents communication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale (TKS) | up to 24 hours post-surgery (0-1 day)
  The kinesiophobia levels of the patients were evaluated postoperatively and 24 hours after surgery.
Pain Level | up to 24 hours post-surgery (0-1 day)
  The pain levels of the patients were measured by means of the visual pain scale.

CONTACTS AND LOCATIONS:
Overall Officials: Gürkan Kapikiran, Ph.D, Principal Investigator — Malatya Turgut Ozal University
Locations (1):
- Turgut Ozal Medical Center, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saritas S, Genc H, Okutan S, Inci R, Ozdemir A, Kizilkaya G. The Effect of Comedy Films on Postoperative Pain and Anxiety in Surgical Oncology Patients. Complement Med Res. 2019;26(4):231-239. doi: 10.1159/000497234. Epub 2019 Mar 27. PMID 30921794
- [Derived] Cici R, Bulbuloglu S, Kapikiran G. Effect of meditation music and comedy movie interventions on postoperative kinesiophobia and pain in patients undergoing total knee arthroplasty. ANZ J Surg. 2023 Jan;93(1-2):302-309. doi: 10.1111/ans.18209. Epub 2022 Dec 14. PMID 36515211